CLINICAL TRIAL: NCT03715335
Title: Improving the Detection of STIs in the Pediatric Emergency Department: A Pragmatic Trial
Brief Title: Adolescent Sexually Transmitted Infection Screening in the Emergency Department
Acronym: STI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: MedStar Health (Other); Nationwide Children's Hospital (Other); Children's National Research Institute (Other); Children's Hospital of Philadelphia (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); Children's Hospital and Health System Foundation, Wisconsin (Other); Baylor College of Medicine (Other); Children's Hospital Colorado (Other); University of Cincinnati (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jennifer Reed, Professor of Clinical Pediatrics, Attending Physician Division of Emergency Medicine, Children's Hospital Medical Center, Cincinnati
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: CIN001-STI Screening; 1R01HD094213-01A1 (NIH)
Record Dates: First submitted 2018-10-11; First posted 2018-10-23 (Actual); Results first posted 2025-11-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-10

CONDITIONS: Gonorrhea; Chlamydia
Keywords: Screening; Emergency Department; Adolescents; Sexually Transmitted Infections; Sexually Transmitted Diseases; Cost Effectiveness; Pragmatic Trial
MeSH Terms: conditions — Gonorrhea; Chlamydia Infections; Emergencies; Sexually Transmitted Diseases

STUDY DESIGN:
Intervention Model Description: A comparative effectiveness pragmatic trial using a stepped wedge crossover design will be conducted. A stepped wedge design involves the sequential roll-out of an intervention or a sequence of interventions to individuals or sites over multiple time periods. At the end of the study, all sites will have received all interventions, but the order in which sites are enrolled is randomly assigned. Once the final intervention is implemented, that intervention will continue until the end of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Baseline (No Intervention): Current STI screening rates.
- Targeted STI Screening (Active Comparator): Data from the Sexual Health Screen (SHS) will be integrated into the Electronic Health Record (EHR) and will provide Clinical Decision Support (CDS) for GC/CT testing based on SHS-calculated STI risk. Patients will be classified as at high risk for STIs, at risk or low risk if they deny any history of sexual activity. When patients classify as at high risk, clinicians will receive CDS that STI testing is "highly recommended"; when they care for patients who classify as at risk, they will receive CDS that STI testing is "recommended"; when caring for patients who classify as at low risk, they will receive CDS that STI testing "is not necessary at this time." If the clinician chooses to follow the recommendation for screening based on patient's risk assessment, and the patient consents to testing on the tablet device, urine GC/CT testing will be performed.
  Interventions: Other: Targeted STI Screening
- Universally Offered STI Screening (Active Comparator): During the universally offered screening intervention, STI screening will be offered to all eligible adolescents, regardless of risk. All eligible patients will also complete the SHS, will be informed of the CDC GC/CT testing recommendations and then be given the option to decline STI testing using the tablet device. During this phase, the SHS results will not be available to the clinician. STI testing recommendations will be based only on the patient's decision to undergo GC/CT testing. Like the process followed in the targeted screening phase, if the clinician follows the CDS that informs the clinician that the patient agreed to GC/CT screening and consequently orders testing, urine GC/CT testing will be performed.
  Interventions: Other: Universally Offered STI Screening

INTERVENTIONS:
Other: Targeted STI Screening — GC/CT screening will be offered to those who screen at risk or at high risk for STIs.
  Arms: Targeted STI Screening
Other: Universally Offered STI Screening — GC/CT screening will be offered to all patients who meet the age eligibility criteria.
  Arms: Universally Offered STI Screening

SUMMARY:
Sexually transmitted infections (STIs) are highly prevalent among adolescents. Clinical practices related to screening, diagnosis, treatment, and prevention of STIs among adolescents are suboptimal. There is a need to expand our screening programs to nontraditional healthcare settings such as emergency departments (ED) and to determine the most efficient and cost-effective method for providing this screening. The goal of this study is to leverage our recent insights obtained from single center ED-based adolescent GC/CT screening research and apply them across a national pediatric ED research network to determine the most clinically effective and cost-effective screening approach for adolescents when implemented into a real-world clinical setting through a pragmatic trial. This will be accomplished through a network of children's hospital EDs with a track record of robust research collaboration (Pediatric Emergency Care Applied Research Network or PECARN). This intervention will rely on an innovative approach that electronically integrates patient-reported data to guide clinical decision support. The investigators will apply human factors modeling methods to perform ED workflow evaluations at each participating pediatric ED to determine the most efficient way to integrate the screening process into clinical care. The investigators will then conduct a comparative effectiveness pragmatic trial of targeted STI screening versus universally offered STI screening through electronic integration of patient reported data for provision of clinical decision support. The investigators will develop decision analytic models to evaluate the cost-effectiveness of targeted screening compared to universally offered screening.

DETAILED DESCRIPTION:
Adolescents are disproportionately affected by sexually transmitted infections (STIs). The STI epidemic among youth is a national public health priority and enhanced STI diagnosis, treatment, and reduction in adolescents is needed.

Adolescents frequently access the emergency department (ED) for care. Although the Centers for Disease Control and Prevention (CDC) recommend universal HIV screening in EDs, no recommendations currently exist for gonorrhea and chlamydia (GC/CT) screening. Addressing the effectiveness and integration of ED-based STI screening is critically needed.

Insufficient knowledge of the ideal structure for delivery is a barrier to the implementation of ED-based GC/CT screening. While universally offered screening (offered to all, regardless of risk) may detect a larger number of cases than targeted screening (screening only those disclosing high risk sexual behavior), it is more resource-intensive and may result in more false positive cases. The investigators each studied targeted (Goyal) and universally offered (Reed) ED-based GC/CT screening via electronically entered patient-reported data providing real-time clinical decision support (CDS). They have shown that both strategies are acceptable, feasible, and result in increased STI screening rates; but it is unknown which method is most efficient and cost effective when instituted across a national sample of pediatric EDs.

The scientific premise of this application is to leverage recent insights obtained from single center ED-based adolescent GC/CT screening research and apply them across a national pediatric ED research network to determine the most clinically effective and cost-effective screening when implemented in a real-world clinical setting. To be sustainable, the ideal screening strategy must be easily incorporated into the clinical workflow. Electronic integration of patient-reported data with CDS offers one such solution. The objective of this study is to compare targeted and universally offered STI screening approaches by seamlessly integrating real-time CDS based on electronically obtained patient-reported data into the normal ED workflow. The investigators will execute a multicenter comparative effectiveness pragmatic trial within a national sample of pediatric EDs through the Pediatric Emergency Care Applied Research Network (PECARN).

Specific Aim 1: To compare the effectiveness of usual care, targeted screening and universally offered screening in EDs through a pragmatic trial that applies a human factors systems approach to implement GC/CT screening into routine clinical care.

Specific Aim 2: To determine the most cost-effective approach for GC/CT detection (i.e. usual care, targeted screening, and universally offered screening) in an adolescent ED population.

Study Design:

1. Workflow Evaluations: The investigators will perform ED workflow evaluations to determine how to best integrate new processes into current workflow by applying a human factors workflow process mapping approach. Data from these methods will enable the development of site-specific adaptations for the implementation of electronically enhanced STI screening processes.
2. Pragmatic Trial: The investigators will then conduct a comparative effectiveness pragmatic trial using a stepped wedge crossover design. Sites will be randomized to one of six positions. After collecting baseline data, each site will subsequently be randomized to either start with implementation of a targeted screening intervention (T) or a universally offered screening intervention (U). Each site will then cross-over and implement the opposite strategy. The final intervention will continue until the conclusion of the study.
3. Cost-effectiveness analysis: Even if universal clinical strategies are proven to be effective, the costs of those strategies compared with usual care or more targeted approaches may make them unsustainable. The result of a cost-effectiveness analysis is the incremental cost-effectiveness ratio (ICER). The investigators plan to look at additional cost per STI detected, as well as cost per QALY gained. The investigators will develop decision analytic models to evaluate the cost-effectiveness of universally offered screening compared with targeted screening and "usual care". A simple model will only examine effectiveness in terms of STIs detected. A more complicated model will include short- and long-term consequences of treated and untreated disease. Based on test characteristics from the literature, small numbers of patients may have false positive or false negative results. The investigators will model the financial and clinical consequences of both. Outcomes will be modeled for unscreened patients who later return for treatment of symptomatic disease. Long-term outcomes addressing the sequelae of untreated/undetected STIs and outcomes following successful detection and treatment will be modeled. Data generated from Aim 2 regarding the effectiveness of the two screening strategies in detecting GC/CT, the proportion of identified patients who ultimately receive treatment, and the prevalence ranges of GC and CT in cohorts presenting for ED care at the 6 sites in this study, will be used to inform probabilities in the model. Literature-based estimates will inform other probabilistic events and costs of long-term STI sequelae in the model. Incremental cost-effectiveness ratios will be calculated to determine cost-effectiveness. A key parameter of interest is the background rate of STI. This likely varies between locations and will be a key determinant to the cost-effectiveness of the universally offered screening strategy. The threshold of background STI prevalence above which universally offered screening becomes "very cost-effective" will be calculated. As a result, the cost-effectiveness of the universally offered screening strategy may vary by location in the study, and in real-world use of the screening tool.

Study Procedures:

1. Human Factors Workflow Analyses: Human factors workflow evaluations will occur at each of the 6 participating sites. These observations will be conducted to understand site-specific ED flow differences that may occur with respect to the care of adolescents. Observational data will be collected regarding ED workflow and information exchange using the tool TaskTracker to record clinical workflow and identify common workflow paths.
2. Pragmatic Trial: Once the ideal workflow strategy is identified at each individual site, all participants in both the targeted and universally offered screening phases will use a tablet device to provide electronic informed consent for participation. All participants will complete the previously developed and validated ACASI SHS containing questions regarding their personal sexual health history. The PROs tool will risk-stratify patients for STIs based on their reported sexual experience and/or presence of STI-related symptoms. Using the tablet device, patients will also provide consent for clinician-ordered urine STI testing. This will provide clinicians real-time EHR-integrated decision support for GC/CT testing. The electronic informed consent document will contain information about the study. Reasons for not offering the tablet will be recorded by the ED staff. If adolescents decline study participation, a reason for refusal will also be recorded on the tablet.

   1. Targeted screening: During the targeted screening intervention, data from the SHS will be integrated into the EHR and will provide CDS for GC/CT testing based on SHS-calculated STI risk. Patients will be classified as high risk for STIs if they disclose being sexually active and have the presence of STI-related symptoms or any of the following high risk behaviors: more than 1 sexual partner in the last 3 months, no condom use during last sex, prior history of STI. Patients will be classified as at risk if they disclose being sexually active but do not disclose having any STI-related symptoms or any high-risk sexual behaviors. Patients will be classified as at low risk if they deny any history of sexual activity. When patients classify as high risk, clinicians will receive CDS that STI testing is "highly recommended"; when they care for patients who classify as at risk, they will receive CDS that STI testing is "recommended". If the clinician chooses to follow the recommendation for screening based on patient's risk assessment, and the patient consents to testing on the tablet device, urine GC/CT testing will be performed.
   2. Universally offered screening: During the universally offered screening intervention, STI screening will be offered to all eligible adolescents, regardless of risk. All eligible patients will also complete the SHS, will be informed of the CDC GC/CT testing recommendations and be given the option to decline STI testing using the tablet device. During this phase, the SHS results will not be available to the clinician. STI testing recommendations will be based only on the patient's decision to undergo GC/CT testing. Like the process followed in the targeted screening phase, if the clinician follows the CDS that informs the clinician that the patient agreed to GC/CT screening and consequently orders testing, urine GC/CT testing will be performed.
   3. Both approaches: If the patient is at risk for STIs and declines GC/CT testing, or the patient simply declines GC/CT testing on the tablet but the clinician believes the patient should be tested, the clinician will have the opportunity to engage in a shared decision-making process with the patient as per routine clinical care. Alternatively, if the clinician declines the CDS GC/CT testing recommendations, he/she will be asked to electronically document the reason the CDS is not being followed. All patients who test positive will be notified of their results and provided treatment based on each site's standard clinical processes for result notification and treatment.

ELIGIBILITY:
Inclusion Criteria

* 15-21 years of age

Exclusion Criteria

* unable to understand English
* critically ill
* cognitive impairment or altered mental status
* unable to provide consent for completion of the sexual health screen and STI screening.

Ages: 15 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 98413 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2022-09-25 (Actual); Study Completion 2025-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Reed, MD, MSCE, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (5):
- United States (5):
  - Colorado Children's Hospital, Aurora, Colorado
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - Children's Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reed JL, Palmer CA, Casper TC, Augustine EM, Cruz AT, Elsholz CL, Mollen CJ, Pickett ML, Schmidt SK, Stukus KS, Goyal MK. Gonorrhea and Chlamydia Screening for Adolescents and Young Adults in Emergency Departments. JAMA Pediatr. 2025 Dec 1;179(12):1343-1352. doi: 10.1001/jamapediatrics.2025.2139. PMID 40920405

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at 6 pediatric emergency departments between January 2021 and September 2023.
Pre-assignment Details: The initial 2-week ramp up period within each screening strategy phase was excluded from all analyses.
Units Other Than Participants: Site
Groups:
- Site A: Sequence 1: 14 weeks of Baseline, 2 weeks of Ramp-Up, 26 weeks of Universally Offered STI Screening, 43 weeks of Targeted STI Screening
- Site B: Sequence 2: 12 weeks of Baseline, 2 weeks of Ramp-Up, 26 weeks of Targeted STI Screening, 45 weeks of Universally Offered STI Screening
- Site C: Sequence 3: 24 weeks of Baseline, 37 weeks of Universally Offered STI Screening, 2 weeks of Ramp-Up, 22 weeks of Targeted STI Screening
- Site D: Sequence 4: 19 weeks Baseline, 2 weeks Ramp-up, 30 weeks Targeted STI Screening, 2 weeks Ramp-up, 32 weeks Universally Offered STI Screening
- Site E: Sequence 5: 17 weeks Baseline, 2 weeks Ramp-up, 26 weeks Universally Offered STI Screening, 2 weeks Ramp-up, 38 weeks Targeted STI Screening
- Site F: Sequence 6: 22 weeks Baseline, 2 weeks Ramp-up, 31 weeks Targeted STI Screening, 30 weeks Universally Offered STI Screening
Period: Overall Study Total
Arm/Group | Site A | Site B | Site C | Site D | Site E | Site F
Started | 24765; 1 Site | 18080; 1 Site | 10969; 1 Site | 23333; 1 Site | 12748; 1 Site | 13144; 1 Site
Completed | 23730; 1 Site | 17200; 1 Site | 10488; 1 Site | 22294; 1 Site | 12153; 1 Site | 12548; 1 Site
Not Completed | 1035; 0 Site | 880; 0 Site | 481; 0 Site | 1039; 0 Site | 595; 0 Site | 596; 0 Site
Period: Baseline
Arm/Group | Site A | Site B | Site C | Site D | Site E | Site F
Started | 3110; 1 Site | 1999; 1 Site | 2753; 1 Site | 5291; 1 Site | 2164; 1 Site | 3316; 1 Site
Completed | 3110; 1 Site | 1999; 1 Site | 2753; 1 Site | 5291; 1 Site | 2164; 1 Site | 3316; 1 Site
Not Completed | 0; 0 Site | 0; 0 Site | 0; 0 Site | 0; 0 Site | 0; 0 Site | 0; 0 Site
Period: Ramp-up 1
Arm/Group | Site A | Site B | Site C | Site D | Site E | Site F
Started | 544; 1 Site | 439; 1 Site | 242; 1 Site | 499; 1 Site | 311; 1 Site | 251; 1 Site
Completed | 544; 1 Site | 439; 1 Site | 242; 1 Site | 499; 1 Site | 311; 1 Site | 251; 1 Site
Not Completed | 0; 0 Site | 0; 0 Site | 0; 0 Site | 0; 0 Site | 0; 0 Site | 0; 0 Site
Period: Screening Intervention 1
Arm/Group | Site A | Site B | Site C | Site D | Site E | Site F
Started | 7732; 1 Site | 5815; 1 Site | 4907; 1 Site | 9252; 1 Site | 4663; 1 Site | 4973; 1 Site
Completed | 7732; 1 Site | 5815; 1 Site | 4907; 1 Site | 9252; 1 Site | 4663; 1 Site | 4973; 1 Site
Not Completed | 0; 0 Site | 0; 0 Site | 0; 0 Site | 0; 0 Site | 0; 0 Site | 0; 0 Site
Period: Ramp-up 2
Arm/Group | Site A | Site B | Site C | Site D | Site E | Site F
Started | 491; 1 Site | 441; 1 Site | 239; 1 Site | 540; 1 Site | 284; 1 Site | 345; 1 Site
Completed | 491; 1 Site | 441; 1 Site | 239; 1 Site | 540; 1 Site | 284; 1 Site | 345; 1 Site
Not Completed | 0; 0 Site | 0; 0 Site | 0; 0 Site | 0; 0 Site | 0; 0 Site | 0; 0 Site
Period: Screening Intervention 2
Arm/Group | Site A | Site B | Site C | Site D | Site E | Site F
Started | 12888; 1 Site | 9386; 1 Site | 2828; 1 Site | 7751; 1 Site | 5326; 1 Site | 4259; 1 Site
Completed | 12888; 1 Site | 9386; 1 Site | 2828; 1 Site | 7751; 1 Site | 5326; 1 Site | 4259; 1 Site
Not Completed | 0; 0 Site | 0; 0 Site | 0; 0 Site | 0; 0 Site | 0; 0 Site | 0; 0 Site

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Targeted STI Screening | Baseline | Universally Offered STI Screening | Total
Number analyzed (Participants) | 41082 | 18633 | 38698 | 98413
Age, Customized [Count of Participants; unit: Participants] — Age at arrival date included <16 years, 16- <18 years, 18- <22 years
  Participants
    Number of Participants: < 16 years of age | 11350 | 5225 | 10774 | 27349
    Number of Participants: 16 - <18 years of age | 21484 | 9573 | 19870 | 50927
    Number of Participants: 18 - < 22 years of age | 8248 | 3835 | 8054 | 20137
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9505 | 4750 | 11368 | 25623
  Not Hispanic or Latino | 27472 | 12368 | 22663 | 62503
  Unknown or Not Reported | 4105 | 1515 | 4667 | 10287
Insurance Status [Count of Participants; unit: Participants]
  Government | 21959 | 9353 | 22052 | 53364
  Commercial | 17500 | 8409 | 14165 | 40074
  Other | 1581 | 867 | 2454 | 4902
  Unknown or Missing | 42 | 4 | 27 | 73
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 23510 | 11037 | 22466 | 57013
  Male | 17532 | 7568 | 16155 | 41255
  Other | 27 | 20 | 56 | 103
  Unknown/Missing | 13 | 8 | 21 | 42
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 13536 | 5606 | 11708 | 30850
  White | 19235 | 9462 | 15814 | 44511
  American Indian/Alaskan Native | 98 | 44 | 124 | 266
  Asian/Pacific Islander | 1038 | 414 | 953 | 2405
  More than one race | 714 | 208 | 677 | 1599
  Other | 5564 | 2522 | 7026 | 15112
  Missing/Unknown | 897 | 377 | 2396 | 3670

OUTCOME MEASURES:

1. Primary Outcome: GC/CT Detection Rates
Description: Our primary outcome measure is GC/CT detection rates per 1000 eligible patients.
Time Frame: Through study completion, an average of 2 years
Population: Patients tested for STI
Measure: Median (Inter-Quartile Range); unit: No. of patients with positive GC/CT
Arm/Group | Baseline | Targeted STI Screening | Universally Offered STI Screening
Number analyzed (Participants) | 1422 | 3023 | 2822
No. of patients with positive GC/CT | 15.2 [12.7 to 17.9] | 12.1 [9.5 to 14.8] | 11 [9.3 to 13.6]

ADVERSE EVENTS:
Time Frame: Adverse data was collected for 798 days
Arm/Group | Baseline | Targeted STI Screening | Universally Offered STI Screening
All-Cause Mortality (participants affected / at risk) | 0/18633 | 0/41082 | 0/38698
Serious Adverse Events (participants affected / at risk) | 0/18633 | 0/41082 | 0/38698
Other Adverse Events (participants affected / at risk) | 0/18633 | 0/41082 | 0/38698

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/35/NCT03715335/Prot_SAP_000.pdf